CLINICAL TRIAL: NCT04940520
Title: Alpha-bisabolol for Onychomycosis Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Adriana Rodrigues dos Anjos Mendonça, Principal Investigator, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Onicomicose
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Onychomycosis
Keywords: Onychomycosis; Phytotherapy; Laser Therapy; Plant Oils
MeSH Terms: conditions — Onychomycosis | interventions — Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Group A: control group, drug recommended by the Brazilian Society of Dermatology
  Interventions: Biological: Drug recommended by the Brazilian Society of Dermatology
- Alpha-bisabolol and laser (Active Comparator): Group B: alpha bisabolol-based product associated with low-level laser therapy
  Interventions: Combination Product: Alpha bisabolol product and laser
- Alpha bisabolol (Active Comparator): Group C: alpha bisabolol based product
  Interventions: Biological: Alpha bisabolol product

INTERVENTIONS:
Biological: Drug recommended by the Brazilian Society of Dermatology — Using a drug recommended by the Brazilian Society of Dermatology, twice a day.
  Arms: Control group
Combination Product: Alpha bisabolol product and laser — Using alpha bisabolol-based product associated with low-level laser therapy. Alpha bisabolol-based product will be used twice a day, and laser therapy used once every fortnight.
  Arms: Alpha-bisabolol and laser
Biological: Alpha bisabolol product — Using alpha bisabolol-based product twice a day
  Arms: Alpha bisabolol

SUMMARY:
Clinical, interventional, longitudinal study with random sampling. 60 patients will be divided into three groups, group A: control group, drug recommended by the Brazilian Society of Dermatology, group B: alpha bisabolol-based product associated with low-level laser therapy, and group C: alpha bisabolol based product. The topical application will be performed twice a day, while the laser application and photographs of the lesions, every 15 days. Areas of the lesions will be compared.

DETAILED DESCRIPTION:
Introduction: Onychomycosis is an infection caused by fungi that feed on keratin, a protein that makes up most of the nails. In patients with diabetes mellitus and onychomycosis, the risk of foot complications is a concern, especially for those who do not perform the practice of self-care of the skin, nails and feet in general correctly, which can trigger an important tissue damage that culminates in limb amputation. One of the alternatives for the treatment are herbal medicines. The application of alpha-bisabolol in the pharmaceutical sector is related to its anti-inflammatory, antispasmodic, antiallergic, drug permeation and deworming properties, having an important action in the morphology of dermatophytic fungal cells. Objectives: Develop and evaluate a pharmaceutical formula with alpha-bisololol for the treatment of onychomycosis. Methods: Clinical, interventional, longitudinal study with random sampling. The study will be held at the Sthomatherapy Clinic of the Nursing Care and Teaching Center at the Samuel Libânio Hospital and at the DermatoCare Clinic Stomatherapy and Podiatry Clinic, Pouso Alegre, MG. 60 patients with onychomycosis will participate in this study, which will be divided into three groups, group A: control group, drug recommended by the Brazilian Society of Dermatology, group B: alpha bisabolol-based product associated with low-level laser therapy, and group C: alpha bisabolol based product. The topical application will be performed twice a day, while the laser application and photographs of the lesions, every 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers with onychomycosis,
* aged over 18 years.

Exclusion Criteria:

* Volunteers have a known allergic process to topical treatment, and those who present an allergic reaction to alpha bisabolol
* patients with a history of neoplasm in a location close to the nail plate, and patients with psoriasis.
* Volunteers who withdraw their consent at any time during the research, and those who present an allergic reaction to alpha bisabolol
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Injury area analysis | 2 months
  All participants will have their nails photographed every 15 days for treatment control and evolution. Theses areas will be compared using the Image J program.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R dos Anjos Mendonça, PhD, Principal Investigator — Vale do Sapucaí University
Locations (1):
- Vale do Sapucaí University, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No